CLINICAL TRIAL: NCT04783857
Title: Modifying Progesterone and Estradiol Levels to Prevent Postpartum Cigarette Smoking Relapse and Reduce Secondhand Smoke Exposure in Infants and Children
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMCH-2021-29672; R01HD100418 (NIH)
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Smoking; Smoking Cessation; Smoking Reduction
MeSH Terms: conditions — Smoking; Smoking Cessation; Smoking Reduction | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Participants in this group will receive progesterone
  Interventions: Drug: Progesterone 200 MG Oral Capsule
- Group 2 (No Intervention): Participants in this group will not receive progesterone

INTERVENTIONS:
Drug: Progesterone 200 MG Oral Capsule — Progesterone, 200mg, once daily, oral tablet/capsule
  Arms: Group 1

SUMMARY:
The investigators aim to address the following specific aims:

* Determine the efficacy of Prog in preventing postpartum smoking relapse and reducing smoking relapse risk factors.
* Examine the effects of this maternal smoking intervention on infant health.
* Examine racial and ethnic differences in intervention outcomes.

DETAILED DESCRIPTION:
This Good Clinical Practice clinical trial will be implemented by an experienced, transdisciplinary, and productive team of investigators to enhance the diversity of the study sample and generalizability of results. We will enroll healthy pregnant women (following enrollment, all subsequent study procedures will be completed postpartum) or postpartum women on hormonal birth control or no hormonal birth control with either a recent history of smoking and a desire to remain abstinent after childbirth, or who are currently smoking and motivated to quit smoking. Participants will be recruited throughout the continental United States (US) and will participant in an observational arm of the study. Participants living in Minnesota (our clinical site) will receive a 12-week course of exogenous progesterone. All participants will be followed for six months with remote visits, self-administered surveys, and self-collection of dried blood spots to measure hormones and smoking-related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent,
* Aged 18 to 45 years old
* Self-reported stable physical and mental health

  1. self-report uncomplicated pregnancy at gestational week 30 or beyond, or
  2. self-report the birth of a child within the past 6 months
* History of ≥ 4 cigarettes per month during the six months prior to pregnancy
* At enrollment, self-report of motivation to become and/or remain abstinent after delivery ≥ 6 on a 10 point Likert-type scale
* Willingness to protect against pregnancy following day 0 to week 12 of the study
* Participants must live in the continental US and have a device to fully participate in the protocol

Exclusion Criteria:

* Current daily use of nicotine replacement therapy or smoking cessation medications, with the exception of e-cigarettes
* Current major depressive disorder based on the Patient Health Questionnaire-9 (PHQ-9) and the Beck Depression Inventory
* Contraindication to progesterone treatment (e.g., current use of drugs that may inhibit CYP3A4; current or history of deep vein thrombosis, pulmonary embolus, clotting or bleeding disorder, hypertension, stroke, heart disease, or liver dysfunction or disease; or peanut allergy),
* Current or within the past 3 months treatment for illicit drug use or alcohol use
* Any condition or issue that, in the opinion of the clinical team, precludes participation in the trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 279 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Smoking abstinence at Month 6 | 6 months
Child health assessed as smoke exposure and acute infant health. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Allen, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Abdelwahab N, Allen A, Harrison K, Petersen A, Allen S. A protocol for modifying progesterone to increase postpartum cigarette smoking abstinence and reduce secondhand smoke exposure in infants. Contemp Clin Trials Commun. 2024 Nov 6;42:101389. doi: 10.1016/j.conctc.2024.101389. eCollection 2024 Dec. PMID 39618477